CLINICAL TRIAL: NCT05355545
Title: Virtually Supervised Exercise for Kidney Transplant Candidates
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Christine Liu, Assistant Professor of Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 65020; 1R01DK133509-01 (NIH)
Record Dates: First submitted 2022-04-22; First posted 2022-05-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Physical Disability

STUDY DESIGN:
Intervention Model Description: This study uses a parallel group delayed intervention design. In the first half of the study (Weeks 0 to 12), the intervention arm will receive the virtually supervised exercise intervention, while the active comparator arm will receive the health education program. In the second half of the study (Weeks 13 to 24), the intervention arm will continue the virtually supervised exercise intervention, while the active comparator group will start the virtually supervised exercise intervention. The primary timepoint of interest will be at 12 weeks.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Virtually supervised exercise (Experimental): In the first half of the study (weeks 0 to 12), participants will receive a virtually supervised exercise program. In the second half of the study (weeks 13 to 24), participant will continue to receive the virtually supervised exercise program.
  Interventions: Behavioral: Virtually supervised exercise
- Health education (Active Comparator): In the first half of the study (weeks 0 to 12), participants will receive a health education program. In the second half of the study (weeks 13 to 24), participant will receive a the virtually supervised exercise program.
  Interventions: Behavioral: Virtually supervised exercise; Behavioral: Health education

INTERVENTIONS:
Behavioral: Virtually supervised exercise — Participants will participate twice weekly in an live exercise program that they will access through a computer connected to the Internet.
Behavioral: Health education — Participants will first participate in a once weekly live health education class that they will access through a computer connected to the Internet. During the second half of the study, participants will participate twice weekly in an live exercise program that they will access through a computer connected to the Internet.
  Arms: Health education

SUMMARY:
This study is examining whether a virtually supervised exercise program can improve physical function in persons who are awaiting kidney transplant. The investigators will compare the results to a similar group of persons who receive a health education program.

DETAILED DESCRIPTION:
This study is examining if a virtually supervised exercise program can improve physical function in persons awaiting kidney transplant. A double-blind, parallel group randomized controlled clinical trial, this study will enroll 80 persons for 24 weeks. Our primary outcome is performance on the 30 second sit to stand test, and our secondary outcomes are changes in the Fatigue Severity Scale and the Beck Depression Inventory.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* Listed for kidney transplant
* Positive answers (e.g. yes) to one of the following:

  * current difficulty with climbing up 10 stairs,
  * has changed in the past year how they climb 10 stairs
  * current difficulty with walking a 0.5 mile (5-6 blocks)
  * has changed in past year in how they walk 0.5 mile (5-6 blocks)
  * documented performance of 430 meters or less on the six minute walk test in the past 12 months
  * documented performance of 9 points or less on the Short Physical Performance Battery in the past 24 months
  * documented performance of less than 3 points or less on the five times sit to stand test in the past 24 months
* Demonstrated ability to stand up independently from a seated position and then sit back down without using their arms or an assistive device in the past 24 months

Exclusion Criteria:

* Does not speak English or Spanish
* Nursing home resident
* Severe low vision (≥20/200 with corrective lens)
* Severe hearing loss even with use of amplification preventing communication
* Unstable angina or uncontrolled arrhythmia
* Supplemental oxygen therapy
* Myocardial infarction, major heart surgery, stroke, venous thromboembolism, hip fracture, hip or knee replacement in past six months (temporary exclusion)
* ≥ 3 errors on the Six Item Screener

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2026-07-07 (Estimated); Study Completion 2026-07-07 (Estimated)

PRIMARY OUTCOMES:
Change in performance on 30 second sit to stand test | Baseline through week 12
  Number of times that a person can stand up from a sitting position in 30 seconds

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the main results will be made available after deidentification.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available beginning 9 months after publication of the main study results. No end date.
Access Criteria: To gain access, data requestors will need to provide a methodologically sound proposal of the planned research and sign a data use agreement.